CLINICAL TRIAL: NCT06144658
Title: VR-MARS Virtual Reality, Medical Assistance and Rescue for Space
Acronym: VR-MARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de Bretagne Sud (Other)
Responsible Party: Principal Investigator, Dr Seamus Thierry, Medical Doctor, Groupe Hospitalier de Bretagne Sud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ID RCB 2019- A03007- 50
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Instructional Virtual Realities; Weightlessness Simulation; Space Simulation; Patient Simulation; High Fidelity Simulation Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmented Reality Headset Usability (Experimental): In this arm, participants tested the functionality and usability of the headset (a Microsoft Hololens 2 or a Varjor XR3)
  Interventions: Device: Augmented Reality Headset / Hololens 2 or Varjo XR3

INTERVENTIONS:
Device: Augmented Reality Headset / Hololens 2 or Varjo XR3 — Augmented Reality Headset

SUMMARY:
VRMARS is a medical simulation study in microgravity. Healthy volunteers (n=18) test in microgravity the functionnality of an augmented reality headset in which a medical assistance is displayed.

ELIGIBILITY:
Inclusion Criteria:

Healthy male or female volunteers.

* Aged between 18 and 66.
* Not currently pregnant.
* Affiliated to a social security system or, for non-Europeans, holders of a European Health Insurance Card (EHIC).
* Have signed written consent for the study.
* Have passed a standard JAR FCL3 Class 2 (Private Pilot Aptitude) medical examination less than 1 year old.

Exclusion Criteria:

On the day of the flight, before the volunteer boards the plane:

* Flu, digestive symptoms (nausea, vomiting), fever.
* Pregnancy: a urine pregnancy test will be performed on the morning of the flight before boarding.
* Altered mental state (flight anxiety, phobia).
* Failure to attend the safety briefing.

During the flight :

* Non-compliance with basic safety instructions.
* Flight-related side effects: fatigue, motion sickness.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Technical validation of the headset in microgravity | 1 day
  The participant had to report to the invistigators whether the headset functioned under microgravity. Images superimposed on the real environment had to be correctly placed and stable in zero-G
Usability test HARUS / Form | 1 day
  The HARUS (Handheld Augmented Reality Usability Scale) is a questionnaire measuring manipulability -- the ease of handling the HAR system, and comprehensibility -- the ease of understanding the information presented by augmented reality.
NASA-TLX cognitive test | 1 day
  The NASA TLX is a subjective, multidimensional assessment tool that rates perceived workload in order to assess a task, system, or team's effectiveness or other aspects of performance (task loading)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier de Bretagne Sud, Lorient, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Access Criteria: on request